CLINICAL TRIAL: NCT05031234
Title: Evaluation of the Benefit of Non-opioid General Anaesthesia on Postoperative Pain in Laparoscopic Colonic Surgery
Acronym: AGORA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020-A02585-34
Record Dates: First submitted 2021-08-16; First posted 2021-09-01 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Colectomy
MeSH Terms: interventions — Anesthesia; Opiate Alkaloids; Morphine

STUDY DESIGN:
Intervention Model Description: Single-centre prospective randomised study carried out in two parallel groups of patients undergoing laparoscopic colectomy.
  * Group 1: conventional general anaesthesia with morphine
  * Group 2: general anaesthesia without opiates
Who Masked: Participant
Masking Description: The patient does not know which treatment is used for the anesthesia
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group with morphine (Active Comparator): conventional general anaesthesia with morphine
  Interventions: Drug: anaesthesia with morphine
- Group without opiates (Experimental): general anaesthesia without opiates
  Interventions: Drug: anaesthesia without opiates

INTERVENTIONS:
Drug: anaesthesia without opiates — Anaesthesia without opiates for patients undergoing laparoscopic colectomy
  Arms: Group without opiates
Drug: anaesthesia with morphine — anaesthesia with morphine for patients undergoing laparoscopic colectomy
  Arms: Group with morphine

SUMMARY:
Evaluation of the benefit of non-opioid general anaesthesia on postoperative pain in laparoscopic colonic surgery

DETAILED DESCRIPTION:
Single-centre prospective randomised study carried out in two parallel groups of patients undergoing laparoscopic colectomy.

* Group 1: conventional general anaesthesia with morphine
* Group 2: general anaesthesia without opiates

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years of age who has read and signed the consent form for participation in the study
* Patient candidate for laparoscopic colectomy (planned or emergency) with possible conversion to laparotomy

Exclusion Criteria:

* Severe renal failure with baseline clearance<30, hepatic failure with baseline PT<40%, cardiac failure with LVEF<20%.
* Patient under court protection, guardianship or curatorship
* Pregnant or breastfeeding patient
* Patient not affiliated to the French social security system
* Impossible to give the subject informed information and/or to give written informed consent: dementia, psychosis, disturbed consciousness, non-French speaking patient
* Contraindication to anaesthesia or to the administration of one of the products used in the anaesthesia protocol
* Patient participating in another interventional research or in a period of exclusion from a previous research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2020-12-17 (Actual); Primary Completion 2023-02-17 (Actual); Study Completion 2023-02-17 (Actual)

PRIMARY OUTCOMES:
Morphine Use | 48 hours
  All intravenous and oral morphine consumed in the first 48 hours after surgery

SECONDARY OUTCOMES:
Postoperative pain H12 | Hour 12
  Postoperative pain will be reported by the nursing staff on a simple numerical scale graduated from 0 to 10 after questioning the patient, according to the usual procedures of the department.
Postoperative pain H24 | Hour 24
  Postoperative pain will be reported by the nursing staff on a simple numerical scale graduated from 0 to 10 after questioning the patient, according to the usual procedures of the department.
Postoperative pain H36 | Hour 36
  Postoperative pain will be reported by the nursing staff on a simple numerical scale graduated from 0 to 10 after questioning the patient, according to the usual procedures of the department.
Postoperative pain H48 | Hour 48
  Postoperative pain will be reported by the nursing staff on a simple numerical scale graduated from 0 to 10 after questioning the patient, according to the usual procedures of the department.
Postoperative pain D30 | Day 30
  Postoperative pain will be reported by the nursing staff on a simple numerical scale graduated from 0 to 10 after questioning the patient, according to the usual procedures of the department.
Mean arterial pressure | 48 hours
  Mean arterial pressure (MAP) (mmHg)
Mean arterial pressure variability | 48 hours
  MAP variability in percentage
Duration of Mean arterial pressure <65 | 48 hours
  Duration of Mean arterial pressure <65 mmHg (min)
Duration of Mean arterial pressure <55 | 48 hours
  Duration of Mean arterial pressure <65 mmHg (min)
Average heart rate | 48 hours
  Average heart rate
Heart rate variability | 48 hours
  Heart rate variability in percentage
Bradycardia duration < 50 | 48 hours
  Bradycardia duration < 50 (min)
Atropine dose administered | 48 hours
  Atropine dose administered (mg)
Ephedrine dose administered | 48 hours
  Ephedrine dose administered (mg)
Noradrenaline dose administered | 48 hours
  Noradrenaline dose administered (ug)
Neosynephrine dose administered | 48 hours
  Neosynephrine dose administered (ug)
Urapidil dose | 48 hours
  Urapidil dose (mg)
Nicardipine dose | 48 hours
  Nicardipine dose (mg)
Postoperative hypoxemia | 48 hours
  Postoperative hypoxemia (Yes/No)
Consumption of non-morphine drug | Day 90
  Consumption of NSAIDs, nefopam, tramadol, ondansetron and other antiemetics
Assessment of tolerance | Day 90
  All adverse events will be collected and compared between the 2 groups
Assessment of disability | Day 30
  Assessment of disability with the World Health Organization Disability Assessment Schedule (WHODAS2.0)
Assessment of disability | Day 90
  Assessment of disability with the World Health Organization Disability Assessment Schedule (WHODAS2.0). Evolution between Day 30 and Day 90.
Time to extubation, time to resumption of transit, time to onset of first gas, length of stay in ICU and total length of hospital stay | Day 90 at least
  Time to extubation, time to resumption of transit, time to onset of first gas, length of stay in ICU and total length of hospital stay
Immediate postoperative hypoxemia | Day 1
  Immediate postoperative hypoxemia
Oxygen requirement | Day 2
  Oxygen requirement (yes/no at D0, D1, D2)

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Privé Médipôle, Villeurbanne, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Collange V, Berruet JB, Aubrun F, Poiblanc M, Olagne E, Golliet Mercier N, Parent S, Noel P, Devillez S, Perrou M, Ramadan J, Coeckelenbergh S, Joosten A. Opioid free versus opioid sparing strategies for multimodal antinociception during laparoscopic colectomy: a randomised controlled trial. Anaesth Crit Care Pain Med. 2024 Dec;43(6):101436. doi: 10.1016/j.accpm.2024.101436. Epub 2024 Oct 9. PMID 39393528